CLINICAL TRIAL: NCT00848744
Title: A Split-Face, Paired-Comparison, Pilot Study to Evaluate Safety and Efficacy of Two Topical Salicylic Acid 1.0% Creams for Mild to Moderate Acne Vulgaris
Brief Title: Comparison of Two Salicylic Acid Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Amy Paller, Chair of the department of dermatology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AP-011008
Record Dates: First submitted 2008-11-24; First posted 2009-02-20 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- topical salicylic acid 1.0% cream (Experimental)
  Interventions: Drug: Formulation A; Drug: Formulation B

INTERVENTIONS:
Drug: Formulation A — Formulation A will be applied to the randomly-assigned single (left or right) side of the face twice daily.
Drug: Formulation B — Formulation B will be applied to the randomly-assigned single (left or right) side of the face twice daily.

SUMMARY:
This study is a split face, paired-comparison, pilot study of at least 10 subjects to complete. Participants in this study will be patients seen at Children's Memorial Hospital, who are clinically diagnosed with mild to moderate acne vulgaris. Participants will be recruited from one of the clinics, as well as from previous Institutional Review Board (IRB) approved acne studies housed in the Department of Dermatology. All subjects accrued from previous studies have agreed to be contacted for further investigations. Subjects 13 to 35 years of age with mild to moderate acne vulgaris symmetrical in appearance on both sides of the face, and meeting inclusion criteria will be eligible to participate

DETAILED DESCRIPTION:
Acne vulgaris is a follicular disorder occurring in pilosebaceous units in the skin of the face, neck, and upper trunk. These sebaceous follicles have follicular channels and adjacent multiacinar sebaceous glands. In the lubrication process of normal skin, sebum travels through the follicular canal to the skin surface, carrying along with it desquamated cells from follicular epithelium. Acne develops when these specialized follicles undergo pathologic alterations that result in the formation of non-inflammatory lesions (comedones) and inflammatory lesions (papules, pustules, and nodules)1.

The basic cause of acne remains unknown, but its manifestations are thought to be the product of four pathogenic events: 1) increased sebum production fueled by androgenic stimulation in the pubertal period; 2) obstruction of the pilosebaceous unit due to an abnormal keratinization process; 3) proliferation of Propionibacterium acnes, an anaerobic diphtheroid normally residing in pilosebaceous follicles; and 4) inflammation that is mediated both by the action of chemotactic factors and various enzymes, and initiated in part by the interaction of P. acnes with toll-like receptors. Impaction of the pilosebaceous follicle gives rise to the microcomedo that is thought to be the precursor lesion of acne1.

Topical salicylic acid is a common and well-established agent with known keratolytic properties used in the treatment of acne vulgaris. The safety profile for topical salicylic acid has been well delineated. The most common side effects attributed to salicylic acid products include irritation, dryness, scaling, burning and stinging.

Salicylic acid 1.0% creams (Formulation A and Formulation B) will be evaluated to detect any differences in their response for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects who are 13 to 35 years of age.
2. Subjects are in good health and are free of any other facial skin disorders that may interfere with acne study assessments.
3. Subjects have the willingness and ability to understand and provide informed assent/consent to participate in the study and are able to communicate with the investigator. Subjects are willing and able to follow all study directions and to commit to all follow-up visits for the duration of the study. In addition, subjects must be willing to accept the restrictions of the study.
4. A minimum of 5 inflammatory lesions (papules and pustules) on each side of the face, and a minimum of 5 non-inflammatory lesions (open comedones and closed comedones on each side of the face. Lesions should be relatively symmetrical in appearance on both sides of the face. At least one inflammatory lesion should be measured no smaller than 2 mm in diameter and should be visible on each side of the face in images taken with digital imaging station.
5. Ongoing oral medications (other than those specifically for acne) are acceptable provided subjects are on a stable regimen throughout the study and provided the medications are determined likely to not interfere with study assessments.
6. Subjects will not use medicated cosmetics and/or soaps (including soaps containing antibacterial agents such as benzoyl peroxide, keratolytic agents such as salicylic acid, skin fresheners/astringents or aftershave lotions) for the duration of the study.
7. Subjects who agree not use any other acne treatment (including prescription and non-prescription medications) on the test site for the duration of the study.
8. Subjects who agree not to change facial cosmetic products during the study.
9. Subjects who agree to only use sunscreen/sunblock agents that are labeled as non-comedogenic.

Exclusion Criteria:

1. Subjects or parents of subjects who are unable to understand the protocol or to give informed consent/assent.
2. Subjects with mental illness.
3. Subjects with no inflammatory acne.
4. Subjects with any acne cysts or nodules.
5. Subjects with acne conglobata, acne fulminans, secondary acne (e.g. Chloracne, drug-induced acne), or any acne requiring systemic treatment.
6. Subjects with excessive facial hair that may interfere with study assessments.
7. Subjects with other facial skin disorders that may interfere with study assessments.
8. Subjects with a history of skin cancer or actinic keratosis.
9. Subjects who have used tanning devices within one week prior to baseline study visit.
10. Subjects who have applied any topical products (e.g. emollients, sunscreens) or any cosmetics to the face at least one hour prior to study assessments.
11. Use of hormonal oral contraceptives for acne control or for less than 6 months prior to study baseline.
12. Subjects with known allergies, a history of allergy or sensitivity to salicylic acid, or any of the test article components.
13. Subjects using topical or systemic medication within 14 days before the study entry, which could interfere with study assessments. This includes but is not limited to the following: anti-inflammatory drugs (e.g. topical and systemic corticosteroids and systemic antihistamines), anti-acne drugs, topical and oral retinoids, topical antibacterial agents to the face, and any immunosuppressive drugs. Ongoing oral medications not expected to interfere with study assessments are allowed if the subject is on a stable regimen.
14. Subjects who are currently enrolled in another clinical investigation or have been enrolled in an acne trial within a period of 30 days prior to enrollment in this study.
15. Subjects who are pregnant or nursing.
16. Subjects who require electrolysis, waxing, or depilatories on the face during conduct of the study.
17. Subjects viewed by the investigator as not being able to complete the study.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Dennis P West, PhD, Study Director — Northwestern University Department of Dermatology
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Salicylic Acid: Participants used salicylic acid Formulation A and B randomized to opposite sides fo the face.on
Period: Overall Study
Arm/Group | Salicylic Acid
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Salicylic Acid
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Assessment
Description: Difference in physician global assessment between two formulations. We remain blinded as to which formulation, both containing salicylic acid, worked better on patients. Measure is a scale (not an option below). Best was 0 (clear), worst was 4 (severe).
Time Frame: 28 days; The visits include baseline, Day 2, Day 7 (+/- 1) and Day 28 (+/- 3).
Population: Analysis was per protocol. Each subject received formulations A and B randomized to opposite sides of the face.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Formulation B: Participants used salicylic acid Formulation A on either the right or left side of the face.
Arm/Group | Salicylic Acid | Formulation B
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 2.65 (0.41) | 2.6 (0.52)
  Day 2 | 2.55 (0.44) | 2.45 (0.55)
  Day 7 | 2.4 (0.61) | 2.3 (0.59)
  Day 28 | 2.20 (0.63) | 2.15 (0.58)

2. Secondary Outcome: The Subject's Medication Side Effect Profile Will be Assessed Using a Application Site Scale for Dryness, Scaling, Redness, and Stinging/Burning.
Time Frame: 4 Weeks
Population: Data were not collected.
Arm/Group | Salicylic Acid | Formulation B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Salicylic Acid
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salicylic Acid (N=10)
irritation and swelling of face (Skin and subcutaneous tissue disorders) | 1 (1) — Subject reported irritation and swelling on the 25th day of study drug use. The symptoms improved after she stopped the study drug within 2 days. She resumed use of study drug and no further reactions were noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No